CLINICAL TRIAL: NCT02740283
Title: The Early Diagnosis of Gestational Diabetes Mellitus Study
Acronym: EDoGDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Bin Liu, Dr., First Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SYSU5010-2016014
Record Dates: First submitted 2016-04-02; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational Diabetes Mellitus; Oral Glucose Tolerance Test
MeSH Terms: conditions — Diabetes, Gestational

ARMS (1):
- Pregnant women (Experimental): As a diagnostic study, the cohort will recruit 300 pregnant women who meet inclusion and exclusion criteria outlined below. OGTTs will be performed between 18 and 20 gestational weeks (early-OGTT) and 24 to 28 gestational weeks (regular-OGTT). Clinical and laboratory information of the mother and their offspring will be collected for analysis.
  Interventions: Behavioral: glycemic monitoring; Dietary Supplement: dietary guide

INTERVENTIONS:
Behavioral: glycemic monitoring
Dietary Supplement: dietary guide

SUMMARY:
The main purpose of the study is to evaluate an OGTT at 18 to 20 gestational weeks as an early diagnosis method of GDM in low risk pregnant women. By investigating maternal and neonatal outcomes that are associated with the early OGTT and regular OGTT results, the study will provide a evidence for the most appropriate time to perform an OGTT in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnant women will be invited to participate in this study if they are between 18 and 40 years of age, and have had their first prenatal visit in our center before 18 weeks 0 days of gestation.

Exclusion Criteria:

* Previous history of GDM or preexisting DM
* Family history of diabetes mellitus (first degree relative with diabetes or a sister with GDM)
* Body mass index>30 kg/m2
* Previous macrosomia (baby with birth weight >4,000 g) or a history of stillbirth
* Polycystic ovary syndrome
* Medications: corticosteroids, antipsychotics
* Participant not willing to take OGTT twice (at 18-20 gestational weeks and 24-28 gestational weeks), or not willing to have a series of prenatal care visits and deliver in our center.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Rate of GDM diagnosed in 18-20 gestational week. | up to 12 months

REFERENCES:
- [Derived] Liu B, Cai J, Xu Y, Long Y, Deng L, Lin S, Zhang J, Yang J, Zhong L, Luo Y, Zhou Y, Zhang Y, Li Z, Chen H, Wang Z. Early Diagnosed Gestational Diabetes Mellitus Is Associated With Adverse Pregnancy Outcomes: A Prospective Cohort Study. J Clin Endocrinol Metab. 2020 Dec 1;105(12):dgaa633. doi: 10.1210/clinem/dgaa633. PMID 32898218
- [Derived] Liu B, Xu Y, Zhang Y, Cai J, Deng L, Yang J, Zhou Y, Long Y, Zhang J, Wang Z. Early Diagnosis of Gestational Diabetes Mellitus (EDoGDM) study: a protocol for a prospective, longitudinal cohort study. BMJ Open. 2016 Nov 21;6(11):e012315. doi: 10.1136/bmjopen-2016-012315. PMID 27872115